CLINICAL TRIAL: NCT03138096
Title: Safety and Protective Efficacy of Genetically Modified Plasmodium Berghei (Pb(PfCS@UIS4)) Malaria Parasites in Healthy Volunteers
Brief Title: Safety and Protective Efficacy of Pb(PfCS@UIS4)
Acronym: PbVac
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: Havenziekenhuis (Other); Erasmus Medical Center (Other); The PATH Malaria Vaccine Initiative (MVI) (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PbVac
Record Dates: First submitted 2017-04-19; First posted 2017-05-03 (Actual); Results first posted 2021-12-15 (Actual); Last update posted 2022-03-04 (Actual); Status verified 2017-03

CONDITIONS: Malaria,Falciparum; Plasmodium Falciparum; Plasmodium Berghei; Controlled Human Malaria Infection (CHMI)
MeSH Terms: conditions — Malaria, Falciparum

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Group 1 - five Pb(PfCS@UIS4)-infected mosquitoes (Experimental): (Group 1) will be exposed to bites of five Pb(PfCS@UIS4)-infected mosquitoes
  Interventions: Biological: Pb(PfCS@UIS4)-infected mosquitoes
- Group 2 - 25 Pb(PfCS@UIS4)-infected mosquito bites (Experimental): (group 2) will be exposed to 25 Pb(PfCS@UIS4)-infected mosquito bites
  Interventions: Biological: Pb(PfCS@UIS4)-infected mosquitoes
- Group 3 - 75 Pb(PfCS@UIS4)-infected mosquito bites (Experimental): (group 3) will be exposed to 75 Pb(PfCS@UIS4)-infected mosquito bites
  Interventions: Biological: Pb(PfCS@UIS4)-infected mosquitoes; Other: Challenge infection P. falciparum
- Group 4 - Infectivity control group of Phase 1 (Other): Infectivity control group of Phase 1
  Interventions: Other: Challenge infection P. falciparum
- Group 5 - Infectivity control group of Phase 2 (Other): Infectivity control group of Phase 2
  Interventions: Other: Challenge infection P. falciparum

INTERVENTIONS:
Biological: Pb(PfCS@UIS4)-infected mosquitoes — Pb(PfCS@UIS4)-infected mosquitoes
  Arms: Group 1 - five Pb(PfCS@UIS4)-infected mosquitoes; Group 2 - 25 Pb(PfCS@UIS4)-infected mosquito bites; Group 3 - 75 Pb(PfCS@UIS4)-infected mosquito bites
Other: Challenge infection P. falciparum — Challenge infection with bites of five infected Pf mosquitoes
  Arms: Group 3 - 75 Pb(PfCS@UIS4)-infected mosquito bites; Group 4 - Infectivity control group of Phase 1; Group 5 - Infectivity control group of Phase 2

SUMMARY:
In the underlying study, a genetically modified P. berghei parasite is used. P. berghei is one of the four Plasmodium species that causes malaria in rodents. The hypothesis is that immunization of humans with P. berghei will induce a cross-species immune response without the risk of a breakthrough infection. To further increase the potential for protective efficacy, the P. falciparum circumsporozoite (CS)- protein gene has been integrated in the P. berghei parasite, generating a genetically modified P. berghei parasite, abbreviated as Pb(PfCS@UIS4).

ELIGIBILITY:
Inclusion Criteria:

1. Subject is aged ≥ 18 and ≤ 35 years and in good health.
2. Subject has adequate understanding of the procedures of the study and is able and willing (in the investigator's opinion) to comply with all study requirements.
3. Subject is willing to complete an informed consent questionnaire and is able to answer all questions correctly.
4. Subject is able to communicate well with the investigator and is available to attend all study visits, lives in Rotterdam or in proximity to the trial centre (can be on site within 1 hour) or is willing to stay in a hotel close to the trial centre during part of the study (phase 1: from day of immunization to day 12 post-immunization; phase 2: from day of immunization to day 8 post-immunization.
5. The subject will remain within the Netherlands from day -1 until day +28 after immunization during phase 1; from day -1 until day 12 after each immunization during phase 2, and during the challenge period, will not travel to a malaria-endemic area during the study period, and is reachable (24/7) by mobile telephone throughout the entire study period.
6. Subject agrees to their general practitioner being informed and contacted about their participation in the study and agrees to sign a form to request the release by their General Practitioner (GP), and medical specialist when necessary, to the investigator(s), of any relevant medical information concerning possible contra-indications for participation in the study.
7. The subject agrees to refrain from blood donation to Sanquin or for other purposes throughout the study period and for a defined period thereafter according to current Sanquin guidelines (3 years minimum, depending on serology).
8. For female subjects: subject agrees to use continuous adequate contraception** and not to breastfeed for the duration of study.
9. Subject agrees to refrain from intensive physical exercise (disproportionate to the subject's usual daily activity or exercise routine) during the malaria challenge period.
10. Subject agrees to avoid additional triggers that may cause elevations in liver enzymes including alcohol from baseline up to 1 week post treatment.
11. Subject has signed written informed consent to participate in the trial.

Exclusion Criteria:

A potential subject who meets any of the following criteria will be excluded from participation in this study:

1. Any history, or evidence at screening, of clinically significant symptoms, physical signs or abnormal laboratory values suggestive of systemic conditions, such as cardiovascular, pulmonary, renal, hepatic, neurological, dermatological, endocrine, malignant, haematological, infectious, immunodeficient, psychiatric and other disorders, which could compromise the health of the volunteer during the study or interfere with the interpretation of the study results. These include, but are not limited to, any of the following.

   1.1. Body weight <50 kg or Body Mass Index (BMI) <18 or >30 kg/m2 at screening. 1.2. A heightened risk of cardiovascular disease, as determined by: an estimated ten year risk of fatal cardiovascular disease of ≥5% at screening, as determined by the Systematic Coronary Risk Evaluation (SCORE); history, or evidence at screening, of clinically significant arrhythmia's, prolonged QT-interval or other clinically relevant ECG abnormalities; or a positive family history of cardiac events in 1st or 2nd degree relatives <50 years old.

   1.3. A medical history of functional asplenia, sickle cell trait/disease, thalassaemia trait/disease or G6PD-deficiency.

   1.4. History of epilepsy in the period of five years prior to study onset, even if no longer on medication.

   1.5. Screening tests positive for Human Immunodeficiency Virus (HIV), active Hepatitis B Virus (HBV), Hepatitis C Virus (HCV) 1.6. Chronic use of i) immunosuppressive drugs, ii) antibiotics, iii) or other immune modifying drugs within three months prior to study onset (inhaled and topical corticosteroids and oral anti-histamines exempted) or expected use of such during the study period.

   1.7. Any recent or current systemic therapy with an antibiotic or drug with potential anti-malarial activity (chloroquine, atovaquone-proguanil, arthemether-lumefantrine, sulfadoxine-pyrimethamine, doxycycline, tetracycline, piperaquine, benzodiazepine, flunarizine, fluoxetine, tetracycline, azithromycin, clindamycin, erythromycin, hydroxychloroquine, etc.) (allowable timeframe for use at the Investigator's discretion).

   1.8. History of malignancy of any organ system (other than localized basal cell carcinoma of the skin), treated or untreated, within the past 5 years.

   1.9. Any history of treatment for severe psychiatric disease by a psychiatrist in the past year.

   1.10. History of drug or alcohol abuse interfering with normal social function in the period of one year prior to study onset, positive urine toxicology test for cocaine or amphetamines at screening or at inclusion, or positive urine toxicology test for cannabis at inclusion.
2. For female subjects: positive urine pregnancy test at screening and/or at the baseline visits, including baseline of immunizations (I-1) and or baseline before CHMI (C-1).
3. Any history of malaria, positive serology for P. falciparum, or previous participation in any malaria (vaccine) study.
4. Known hypersensitivity to or contra-indications (including co-medication) for use of sulfadoxine-pyrimethamine, piperaquine, chloroquine, Malarone®, artemether-lumefantrine, primaquine or history of severe (allergic) reactions to mosquito bites.
5. Receipt of any vaccinations in the 3 months prior to the start of the study or plans to receive any other vaccinations during the study period or up to 8 weeks thereafter.
6. Participation in any other clinical study in the 30 days prior to the start of the study or during the study period.
7. Being an employee or student of the department of Medical Microbiology and Infectious Diseases of the Erasmus MC or Radboudumc, or the department of Internal Medicine of the Radboudumc or Havenziekenhuis.
8. Any other condition or situation that would, in the opinion of the investigator, place the subject at an unacceptable risk of injury or render the subject unable to meet the requirements of the protocol.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2017-05-29 (Actual); Primary Completion 2018-03-28 (Actual); Study Completion 2018-10-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Sauerwein, MD PhD, Principal Investigator — Radboud University Medical Center
Locations (2):
- Netherlands (2):
  - Radboud university medical center, Nijmegen, Gelderland
  - Havenziekenhuis, Rotterdam

IPD SHARING:
Plan to Share IPD: Yes
Results will be published

REFERENCES:
- [Result] Reuling IJ, Mendes AM, de Jong GM, Fabra-Garcia A, Nunes-Cabaco H, van Gemert GJ, Graumans W, Coffeng LE, de Vlas SJ, Yang ASP, Lee C, Wu Y, Birkett AJ, Ockenhouse CF, Koelewijn R, van Hellemond JJ, van Genderen PJJ, Sauerwein RW, Prudencio M. An open-label phase 1/2a trial of a genetically modified rodent malaria parasite for immunization against Plasmodium falciparum malaria. Sci Transl Med. 2020 May 20;12(544):eaay2578. doi: 10.1126/scitranslmed.aay2578. PMID 32434846

RESULTS

PARTICIPANT FLOW:
Groups:
- Group 3 -25 Pb(PfCS@UIS4)-Infected Mosquito Bites: (group 3) will be exposed to 75 Pb(PfCS@UIS4)-infected mosquito bites
  Pb(PfCS@UIS4)-infected mosquitoes: Pb(PfCS@UIS4)-infected mosquitoes
  Challenge infection P. falciparum: Challenge infection with bites of five infected Pf mosquitoes
- Group 4 - Infectivity Control Group (Phase 1): Infectivity control group (Phase 1)
  Challenge infection P. falciparum: Challenge infection with bites of five infected Pf mosquitoes
- Group 5 - Infectivity Control Group (Phase 2): Infectivity control group of Phase 2
  Challenge infection P. falciparum: Challenge infection with bites of five infected Pf mosquitoes
Period: Overall Study
Arm/Group | Group 1 - Five Pb(PfCS@UIS4)-Infected Mosquitoes | Group 2 - 25 Pb(PfCS@UIS4)-Infected Mosquito Bites | Group 3 -25 Pb(PfCS@UIS4)-Infected Mosquito Bites | Group 4 - Infectivity Control Group (Phase 1) | Group 5 - Infectivity Control Group (Phase 2)
Started | 3 | 3 | 12 | 6 | 0 (Phase 2 was not started because of unsufficient effectivity of the Pb(PfCS@UIS4) immunizations as pre-determined in the study protocol.)
Completed | 3 | 3 | 12 | 6 | 0
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: phase 2 was not effected
Groups:
- Group 1: (Group 1) will be exposed to bites of five Pb(PfCS@UIS4)-infected mosquitoes
  Pb(PfCS@UIS4)-infected mosquitoes: Pb(PfCS@UIS4)-infected mosquitoes
- Group 2: (group 2) will be exposed to 25 Pb(PfCS@UIS4)-infected mosquito bites
  Pb(PfCS@UIS4)-infected mosquitoes: Pb(PfCS@UIS4)-infected mosquitoes
- Group 3: (group 3) will be exposed to 75 Pb(PfCS@UIS4)-infected mosquito bites
  Pb(PfCS@UIS4)-infected mosquitoes: Pb(PfCS@UIS4)-infected mosquitoes
  Challenge infection P. falciparum: Challenge infection with bites of five infected Pf mosquitoes
- Group 4; Group 5: Infectivity control group
  Challenge infection P. falciparum: Challenge infection with bites of five infected Pf mosquitoes
- Total: Total of all reporting groups
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Group 5 | Total
Number analyzed (Participants) | 3 | 3 | 12 | 6 | 0 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 |  | 0
  Between 18 and 65 years | 3 | 3 | 12 | 6 |  | 24
  >=65 years | 0 | 0 | 0 | 0 |  | 0
Age, Continuous [Median (Full Range); unit: Years] | 21.1 [18 to 23] | 26.1 [21 to 30] | 21.5 [19 to 26] | 22.5 [21 to 26] |  | 22.5 [18 to 30]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 7 | 4 |  | 15
  Male | 0 | 2 | 5 | 2 |  | 9
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Netherlands | 3 | 3 | 12 | 6 |  | 24

OUTCOME MEASURES:

1. Primary Outcome: Adverse Events in Study Groups Following Exposure to Pb(PfCS@UIS4)-Infected Mosquitoes [Safety]
Description: Frequency and magnitude of adverse events in study groups following one or more exposures to Pb(PfCS@UIS4)-infected mosquitoes.
Time Frame: Groups 1&2: from exposure to Pb(PfCS@UIS4)-infected mosquitoes until 28 days thereafter. Group 3: from first exposure until 21 days after fourth/final exposure (=until day immediately prior to CHMI, i.e. approximately 15 weeks after first exposure).
Population: Groups 1-3, immunization phase only (groups 1&2 underwent only a single immunization; group 3 underwent 4 sequential immunizations). Note: group 4 did NOT undergo immunization. AEs following CHMI with WT-infected mosquitoes (i.e. in group 3&4) were not a protocol-defined endpoint and are NOT included here. Group 5 was not enrolled, as protective efficacy in group 3 following first CHMI was insufficient (per protocol) to warrant a second CHMI and hence a second infectivity control group.
Measure: Number; unit: numbers of adverse events
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Number analyzed (Participants) | 3 | 3 | 12 | 0
numbers of adverse events
  Immunization 1: Numbers of local adverse events (grade 1/2) | 0 | 3 | 10 |
  Immunization 2: Numbers of local adverse events (grade 1/2): number analyzed (Participants) | 0 | 0 | 12 | 0
  Immunization 2: Numbers of local adverse events (grade 1/2) |  |  | 9 |
  Immunization 3: Numbers of local adverse events (grade 1/2): number analyzed (Participants) | 0 | 0 | 12 | 0
  Immunization 3: Numbers of local adverse events (grade 1/2) |  |  | 12 |
  Immunization 4: Numbers of local adverse events (grade 1/2): number analyzed (Participants) | 0 | 0 | 12 | 0
  Immunization 4: Numbers of local adverse events (grade 1/2) |  |  | 11 |
  Immunization 1: Numbers of systemic adverse events (grade 1/2) | 7 | 5 | 9 |
  Immunization 2: Numbers of systemic adverse events (grade 1/2): number analyzed (Participants) | 0 | 0 | 12 | 0
  Immunization 2: Numbers of systemic adverse events (grade 1/2) |  |  | 2 |
  Immunization 3: Numbers of systemic adverse events (grade 1/2): number analyzed (Participants) | 0 | 0 | 12 | 0
  Immunization 3: Numbers of systemic adverse events (grade 1/2) |  |  | 4 |
  Immunization 4: Numbers of systemic adverse events (grade 1/2): number analyzed (Participants) | 0 | 0 | 12 | 0
  Immunization 4: Numbers of systemic adverse events (grade 1/2) |  |  | 4 |

2. Primary Outcome: Presence of Breakthrough Parasitemia Following Exposure to Pb(PfCS@UIS4)-Infected Mosquito Bites
Description: Presence of breakthrough parasitemia following (first) exposure to Pb(PfCS@UIS4)-infected mosquito bites, as determined by thick blood smear microscopy
Time Frame: Groups 1-3: from (first) exposure until 28 days thereafter.
Population: Groups 1-3 only. Note: For group 3, only immunisation (exposure) #1 is included here, as immunisations #2-4 fell in phase 2 of the trial, during which this outcome was no longer classified as an endpoint. Group 4 was not exposed to Pb(PfCS@UIS4)-infected mosquitoes (only to CHMI with WT-infected mosquitoes) and group 5 was not enrolled, as protective efficacy in group 3 following first CHMI was insufficient (per protocol) to warrant a second CHMI and hence a second infectivity control group.
Measure: Count of Participants; unit: Participants
Groups:
- Group 1 -Five Pb(PfCS@UIS4)-Infected Mosquitoes: (Group 1) will be exposed to bites of five Pb(PfCS@UIS4)-infected mosquitoes
  Pb(PfCS@UIS4)-infected mosquitoes: Pb(PfCS@UIS4)-infected mosquitoes
- Group 4 - Infectivity Control Group: Infectivity control group
  Challenge infection P. falciparum: Challenge infection with bites of five infected Pf mosquitoes
  No exposure to Pb(PfCS@UIS4)
Arm/Group | Group 1 -Five Pb(PfCS@UIS4)-Infected Mosquitoes | Group 2 - 25 Pb(PfCS@UIS4)-Infected Mosquito Bites | Group 3 - 75 Pb(PfCS@UIS4)-Infected Mosquito Bites | Group 4 - Infectivity Control Group
Number analyzed (Participants) | 3 | 3 | 12 | 0
Participants | 0 | 0 | 0 |

3. Primary Outcome: Time to Parasitemia After CHMI [Efficacy]
Description: Time to parasitemia after CHMI with the wild-type NF54 P. falciparum strain, as detected by qPCR [Efficacy]
Time Frame: Groups 3&4: from day of CHMI until 28 days thereafter
Population: Groups 3&4 only. Note: Groups 1 & 2 did not undergo CHMI and group 5 was not enrolled, as protective efficacy in group 3 following first CHMI was insufficient (per protocol) to warrant a second CHMI and hence a second infectivity control group
Measure: Mean (Full Range); unit: days to P. falciparum parasitemia
Groups:
- Group 1 -Five Pb(PfCS@UIS4)-Infected Mosquitoes: (Group 1) will be exposed to bites of five Pb(PfCS@UIS4)-infected mosquitoes
  Pb(PfCS@UIS4)-infected mosquitoes: Pb(PfCS@UIS4)-infected mosquitoes
  Not exposed to P. falciparum
- Group 2 - 25 Pb(PfCS@UIS4)-Infected Mosquito Bites: (group 2) will be exposed to 25 Pb(PfCS@UIS4)-infected mosquito bites
  Pb(PfCS@UIS4)-infected mosquitoes: Pb(PfCS@UIS4)-infected mosquitoes
  Not exposed to P. falciparum
- Group 4 - Infectivity Control Group: Infectivity control group
  Challenge infection P. falciparum: Challenge infection with bites of five infected Pf mosquitoes
Arm/Group | Group 1 -Five Pb(PfCS@UIS4)-Infected Mosquitoes | Group 2 - 25 Pb(PfCS@UIS4)-Infected Mosquito Bites | Group 3 - 75 Pb(PfCS@UIS4)-Infected Mosquito Bites | Group 4 - Infectivity Control Group
Number analyzed (Participants) | 0 | 0 | 12 | 6
days to P. falciparum parasitemia |  |  | 9.9 [7 to 14] | 7.7 [7 to 11]

4. Secondary Outcome: Immunogenicity of Pb(PfCS@UIS4) as Assessed by ELISA
Description: Immunogenicity of repeated Pb(PfCS@UIS4) immunization as assessed by fold change in anti-P. falciparum IgG from baseline to post-immunization (day prior to CHMI), as measured by ELISA.
Time Frame: Group 3: from baseline until day prior to CHMI (approximately 15 weeks after first Pb(PfCS@UIS4) immunization)
Population: Group 3 only. Note: no analysis of humoral immune responses was performed for Groups 1 & 2 (single immunization only) or group 4 (no immunization); group 5 was not enrolled.
Measure: Mean (Standard Deviation); unit: Fold increase in anti-P. falciparum IgG
Groups:
- Group 1: (Group 1) will be exposed to bites of five Pb(PfCS@UIS4)-infected mosquitoes
  Pb(PfCS@UIS4)-infected mosquitoes: Pb(PfCS@UIS4)-infected mosquitoes
  No humoral responses measured
- Group 2: (group 2) will be exposed to 25 Pb(PfCS@UIS4)-infected mosquito bites
  Pb(PfCS@UIS4)-infected mosquitoes: Pb(PfCS@UIS4)-infected mosquitoes
  No humoral responses measured
- Group 4: Infectivity control group
  Challenge infection P. falciparum: Challenge infection with bites of five infected Pf mosquitoes
  No humoral responses measured
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Number analyzed (Participants) | 0 | 0 | 12 | 0
Fold increase in anti-P. falciparum IgG |  |  | 3.5 (0.3) |

5. Other Pre Specified Outcome: Cellular Immune Responses After Exposure to Pb(PfCS@UIS4) [Exploratory Endpoint]
Description: Cellular immune responses after repeated exposure to Pb(PfCS@UIS4), as determined by increase in %-age IFNg+ lymphocytes following in vitro stimulation of PBMCs with WT P. falciparum sporozoites measured by flow cytometry at baseline and following immunization (day prior to CHMI)
Time Frame: Group 3: from baseline until day prior to CHMI (approximately 15 weeks after first Pb(PfCS@UIS4) immunization)
Population: Group 3 only. Note: no analysis of cellular immune responses was performed for Groups 1 & 2 (single immunization only) or group 4 (no immunizsation); group 5 was not enrolled.
Measure: Mean (Standard Deviation); unit: change in %-age IFNg+ lymphocytes
Arm/Group | Group 1 - Five Pb(PfCS@UIS4)-Infected Mosquitoes | Group 2 - 25 Pb(PfCS@UIS4)-Infected Mosquito Bites | Group 3 - 75 Pb(PfCS@UIS4)-Infected Mosquito Bites | Group 4 - Infectivity Control Group
Number analyzed (Participants) | 0 | 0 | 12 | 0
change in %-age IFNg+ lymphocytes |  |  | 0.510 (1.102) |

6. Other Pre Specified Outcome: Humoral Immune Responses After Exposure to Pb(PfCS@UIS4) [Exploratory Endpoint]
Description: Humoral immune responses after repeated exposure to Pb(PfCS@UIS4) as determined by increase in %-age inhibition of WT P. falciparum sporozoite invasion in HC-04 cells by purified plasma IgG collected at baseline and following immunization (day prior to CHMI).
Time Frame: Group 3: from baseline until day prior to CHMI (approximately 15 weeks after first Pb(PfCS@UIS4) immunization)
Population: Group 3 only. Note: no analysis of humoral immune responses was performed for Groups 1 & 2 (single immunizsation only) or group 4 (no immunization); group 5 was not enrolled.
Measure: Mean (Standard Deviation); unit: % change in inhibition of spz invasion
Groups:
- Group 1 - Five Pb(PfCS@UIS4)-Infected Mosquitoes: (Group 1) will be exposed to bites of five Pb(PfCS@UIS4)-infected mosquitoes
  Pb(PfCS@UIS4)-infected mosquitoes: Pb(PfCS@UIS4)-infected mosquitoes
  No humoral responses measured
- Group 2 - 25 Pb(PfCS@UIS4)-Infected Mosquito Bites: (group 2) will be exposed to 25 Pb(PfCS@UIS4)-infected mosquito bites
  Pb(PfCS@UIS4)-infected mosquitoes: Pb(PfCS@UIS4)-infected mosquitoes
  No humoral responses measured
Arm/Group | Group 1 - Five Pb(PfCS@UIS4)-Infected Mosquitoes | Group 2 - 25 Pb(PfCS@UIS4)-Infected Mosquito Bites | Group 3 - 75 Pb(PfCS@UIS4)-Infected Mosquito Bites | Group 4 - Infectivity Control Group
Number analyzed (Participants) | 0 | 0 | 12 | 0
% change in inhibition of spz invasion |  |  | 48.8 (17.5) |

ADVERSE EVENTS:
Time Frame: 79 days
Description: Blood was drawn for routine haematological and biochemical analysis and peripheral thick blood smears. Signs and symptoms were recorded and graded by a physician. An independent Safety Monitoring Committee was appointed to assess safety data as presented by the study team in periodic safety reports. These reports included comprehensive lists of adverse events and any safety laboratory values outside the normal range.
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3 | 0/12 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3 | 0/12 | 0/6
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 11/12 | 6/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1 (N=3) | Group 2 (N=3) | Group 3 (N=12) | Group 4 (N=6)
Pruritis (Skin and subcutaneous tissue disorders) | 0 | 3 | 10 | 1
Edema arms (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Painful skin arms (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Hematoma / Pain after venapuncture (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1
Headache (General disorders) | 2 | 2 | 7 | 6
Abdominal pain (General disorders) | 1 | 0 | 1 | 0
Nausea (General disorders) | 2 | 0 | 6 | 4
Diarrhoea (General disorders) | 1 | 1 | 1 | 0
Stomach pain (General disorders) | 0 | 1 | 1 | 0
Malaise (General disorders) | 0 | 0 | 4 | 2
Fatigue (General disorders) | 0 | 1 | 4 | 0
Angio-oedema (General disorders) | 0 | 0 | 1 | 0
Dizziness (General disorders) | 1 | 0 | 0 | 0
Night sweating (General disorders) | 0 | 0 | 1 | 0
Chills (General disorders) | 0 | 0 | 1 | 0
Myalgia (General disorders) | 0 | 0 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-11-28): https://cdn.clinicaltrials.gov/large-docs/96/NCT03138096/Prot_SAP_000.pdf